CLINICAL TRIAL: NCT00789802
Title: A Randomized, Controlled Trial of Oral Naproxen and Transdermal Estradiol for Prevention of Unscheduled Bleeding in New Users of Levonorgestrel Intrauterine Contraception
Brief Title: A Randomized Controlled Trial of Oral Naproxen and Transdermal Estradiol for Bleeding in LNG-IUC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other)
Responsible Party: Principal Investigator, Tessa Madden, MD, Asst. Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-1026
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Contraception; Bleeding
Keywords: contraception; progestin contraception; intrauterine contraception; unscheduled bleeding; placebo
MeSH Terms: conditions — Hemorrhage | interventions — Estradiol; Naproxen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- transdermal estradiol (Experimental): participants will be randomized to transdermal estradiol
  Interventions: Drug: transdermal estradiol
- oral naproxen (Experimental): participants will be randomized to oral naproxen
  Interventions: Drug: naproxen
- oral placebo (Placebo Comparator): participants will be randomized to oral placebo
  Interventions: Drug: oral placebo

INTERVENTIONS:
Drug: transdermal estradiol — transdermal estradiol 0.1mg patch to be changed weekly for 12 weeks.
  Other Names: Climara
  Arms: transdermal estradiol
Drug: naproxen — naproxen 500mg by mouth twice daily for the first 5 days of every 4 week period for a total of 12 weeks
  Other Names: Naprosyn, Anaprox
  Arms: oral naproxen
Drug: oral placebo — oral placebo to be taken by mouth twice daily for the first 5 days of a 4 week block for a total of 5 weeks
  Arms: oral placebo

SUMMARY:
We hypothesize that the addition of oral naproxen or transdermal estradiol will decrease the number of days of unscheduled bleeding experienced by first-time users of the levonorgestrel intrauterine system (LNG-IUC) during the first 12 weeks of use compared to an oral placebo. The objective of this study is to compare the total number of days of bleeding experienced by first time users of the LNG-IUC randomized to oral naproxen or estradiol patch compared to those randomized to placebo for the first 12 weeks of use. We will enroll women initiating LNG-IUC to one of 3 groups, transdermal estrogen, oral naproxen or oral placebo. We will enroll a total of 114 women, 38 in each group. Women will keep bleeding diaries for 16 weeks which will be used to calculate the total number of bleeding or spotting days. Statistical analysis will be performed to evaluate if there is less bleeding among the treatment arms then the placebo arm.

DETAILED DESCRIPTION:
The levonorgestrel intrauterine system (LNG-IUC) is one of the most effective, reversible methods of contraception currently available in the United States. User satisfaction is overall high , however the most often cited reason for discontinuation is irregular bleeding . The LNG-IUC has mainly progesteronic effects on the uterine cavity. Morphological changes of the endometrium are observed, including stromal pseudo-decidualization and glandular atrophy . These endometrial changes may contribute to the irregular uterine bleeding experienced by women using the LNG-IUC. Up to 14% of women will discontinue the LNG-IUC within the 5-year period due to abnormal bleeding and up to 66% of woman who request removal of the LNG-IUC will do so in the first 6 months of use . Women may be less likely to discontinue the LNG-IUC due to abnormal bleeding patterns if they are counseled appropriately beforehand, however the prospect of irregular bleeding with few options for management may dissuade some women from even trying the LNG-IUC. A recent Cochrane review identified the need for further investigation into the treatment of irregular uterine bleeding caused by progestin only contraception .

One treatment for progestin-induced irregular bleeding is the administration of nonsteroidal anti-inflammatory agents (NSAIDs). A 1999 study showed a significant decrease in the number of bleeding days in women using the levonorgestrel sub-dermal implant randomized to mefenamic acid 500 mg compared to placebo . A 2004 study found a 50% reduction in bleeding in depot medroxyprogesterone (DPMA) users randomized to mefenamic acid versus placebo . There have been no studies looking specifically at NSAIDs for the prevention or treatment of LNG-IUC related irregular bleeding. Naproxen is an antiprostaglandin that is commonly used in gynecological practice for relief of dysmenorrhea and has been used to treat menorrhagia. It is widely available, inexpensive, well-tolerated and has a low incidence of side effects.

Previous studies have also shown the administration of estrogen alone and estrogen-containing oral contraceptives to users of subdermal levonorgestrel implants (Norplant®) resulted in decreased frequency of irregular uterine bleeding , . A prior randomized, controlled trial found a 0.1mg estradiol patch resulted in the clinical improvement of abnormal bleeding, however this finding was not statistically significant . A randomized, controlled trial of DMPA users found the cyclic administration of 0.1mg estradiol patches did not decreases irregular menstrual bleeding . In this study, the cyclic use of estrogen may have resulted in lower or inconsistent serum estradiol levels. Additionally, the progestational mechanism of action is more similar between levonorgestrel subdermal implants and LNG-IUC than depot medroxyprogesterone. No study has specifically addressed estrogen for treatment of irregular bleeding with the LNG-IUC.

ELIGIBILITY:
Inclusion Criteria:

* Must be of reproductive age from 18 to 45 years
* Must be choosing LNG-IUC for contraception
* Must be English-speaking
* Be willing to avoid additional use of exogenous hormones, such as oral contraceptives, for the duration of the study
* Be willing to avoid additional use of nonsteroidal antiinflammatory drugs, such as ibuprofen or aspirin for the duration of the study
* Be willing to comply with the study protocol, keep the bleeding diary and comply with follow-up visits and telephone interviews as scheduled
* Be willing and able to provide informed consent

Exclusion Criteria:

* Known or suspected pregnancy
* Contraindication to estrogen use, such as presence or history of:

  * venous thromboembolism
  * Arterial thrombosis
  * Thrombophilia disorders, or known family history of
  * Hypertension
  * Migraine headaches with aura or focal neurologic involvement, or any migraine over age 35 years
* Recent or planned future major surgery which will result in prolonged immobilization during the study period
* Presence or history of severe hepatic disease or liver tumors
* Known or suspected estrogen-dependent neoplasm
* Vaginal bleeding of unknown etiology
* Any cigarette smoking and age over 35 years
* Contraindications to nonsteroidal anti-inflammatory use, such as presence or history of:

  * Gastrointestinal ulcer disease
  * Renal insufficiency or failure
  * Aspirin-induced asthma or hypersensitivity reaction
  * Systemic lupus erythematosus (SLE) and mixed connective tissue disorders
  * Use of anticoagulants
  * Cardiovascular disease
* Use of medications that alter estrogen metabolism, i.e. rifampin, certain anti-seizure medications
* Regular use of an NSAID
* Current diagnosis of menorrhagia, metrorrhagia, symptomatic uterine fibroids, or endometrial polyp
* Hypersensitivity or allergy to any of the components of the estradiol patch
* Use of injectable contraception within 6 months of the start of the study medication
* Delivery or abortion in the previous 4 weeks
* Prior use of LNG-IUD
* Any condition, that in the opinion of the investigator, would contraindicate study participation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tessa E Madden, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School fo Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 129 participants were recruited from November 2008 to January 2010 and follow-up was conducted through May 2010.
Groups:
- Oral Naproxen: participants will be randomized to oral naproxen
  naproxen : naproxen 500mg by mouth twice daily for the first 5 days of every 4 week period for a total of 12 weeks
- Oral Placebo: oral placebo : oral placebo to be taken by mouth twice daily for the first 5 days of a 4 week block for a total of 5 weeks
- Transdermal Estradiol: participants will be randomized to transdermal estradiol
  transdermal estradiol : transdermal estradiol 0.1mg patch to be changed weekly for 12 weeks.
Period: Overall Study
Arm/Group | Oral Naproxen | Oral Placebo | Transdermal Estradiol
Started | 44 | 42 | 43
Completed | 34 | 35 | 37
Not Completed | 10 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Naproxen | Oral Placebo | Transdermal Estradiol | Total
Number analyzed (Participants) | 44 | 42 | 43 | 129
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 42 | 43 | 129
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (4.7) | 25 (4.2) | 26.2 (5.1) | 25.8 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 42 | 43 | 129
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 42 | 43 | 129

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding and Spotting Days
Description: The median number of bleeding and spotting days reported at 12 weeks.
Time Frame: 12 weeks
Measure: Median (Full Range); unit: DAYS
Arm/Group | Oral Naproxen | Oral Placebo | Transdermal Estradiol
Number analyzed (Participants) | 44 | 42 | 43
DAYS | 27.5 [5 to 83] | 32 [9 to 84] | 44 [2 to 82]
Statistical Analysis 1: Comparison: Oral Naproxen vs Oral Placebo; Test type: Superiority or Other; p = .03, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oral Placebo vs Transdermal Estradiol; Test type: Superiority or Other; p = .02, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Bleeding Days Observed in Women With a LNG-IUC Treated With Naproxen, Estradiol and Placebo.
Description: Median number of bleeding days observed in women with a LNG-IUC treated with naproxen, estradiol and placebo at 16 weeks.
Time Frame: 16 weeks
Population: There 129 women who were randomly assigned to the 3 arms. At 12 weeks of follow up, there were 17 participants lost to follow up. This resulted in a total analysis population of 112 participants.
Measure: Median (Full Range); unit: days
Arm/Group | Transdermal Estradiol | Oral Naproxen | Oral Placebo
Number analyzed (Participants) | 42 | 44 | 43
days | 35 [11 to 111] | 53 [2 to 106] | 38 [10 to 102]

3. Secondary Outcome: Patient Satisfaction With the LNG-IUC at the End of the 12 Weeks Between the 3 Study Groups.
Description: To compare the level of patient satisfaction with the LNG-IUC at the end of the 12 weeks between the 3 study groups.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Naproxen | Oral Placebo | Transdermal Estradiol
Number analyzed (Participants) | 36 | 39 | 37
Participants
  Satisfied | 26 | 34 | 26
  Somewhat satisfied | 6 | 5 | 6
  Not satisfied | 4 | 0 | 5

4. Secondary Outcome: Continuation Rates of the LNG-IUC at the End of the 12 Week Between the 3 Study Groups
Description: To compare continuation rates of the LNG-IUC at the end of the 12 week between the 3 study groups
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Naproxen | Oral Placebo | Transdermal Estradiol
Number analyzed (Participants) | 44 | 42 | 43
Participants | 34 | 35 | 37

ADVERSE EVENTS:
Arm/Group | Oral Naproxen | Oral Placebo | Transdermal Estradiol
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 0/44 | 0/42 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No